CLINICAL TRIAL: NCT07396519
Title: Bioequivalence Study of Dronedarone Hydrochloride Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NTP-JNDL-T-BEO1
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronedarone Hydrochloride Tablets (Experimental): Healthy male subjects will be randomized to receive a single oral dose of the Test and Reference formulations under fed conditions (30 minutes after a high-fat, high-calorie meal), according to a two-period, two-sequence crossover design with a 10-day washout period between periods.
  Interventions: Drug: Dronedarone Hydrochloride Tablets
- MULTAQ® (Active Comparator): Healthy male subjects will be randomized to receive a single oral dose of the Test and Reference formulations under fed conditions (30 minutes after a high-fat, high-calorie meal), according to a two-period, two-sequence crossover design with a 10-day washout period between periods.
  Interventions: Drug: MULTAQ® (Dronedarone Hydrochloride Tablets)

INTERVENTIONS:
Drug: Dronedarone Hydrochloride Tablets — Test Product. Manufacturer: Shandong New Time Pharmaceutical Co., Ltd. Dosage Form/Strength: 400 mg tablet Administration: Single oral dose of 400 mg (1 tablet).
  Arms: Dronedarone Hydrochloride Tablets
Drug: MULTAQ® (Dronedarone Hydrochloride Tablets) — Reference Product. Manufacturer: Sanofi-Aventis U.S. LLC Dosage Form/Strength: 400 mg tablet Administration: Single oral dose of 400 mg (1 tablet).
  Arms: MULTAQ®

SUMMARY:
The test formulation of Dronedarone Hydrochloride Tablets (400 mg) is bioequivalent to the reference formulation (MULTAQ®) in healthy Chinese subjects under fed conditions.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, single-dose, two-formulation, two-sequence crossover study designed to evaluate the bioequivalence and safety of a generic formulation versus the reference formulation of Dronedarone Hydrochloride Tablets (400 mg) in healthy Chinese male subjects under fed conditions. A planned total of 48 eligible subjects will be enrolled.

Venous blood samples are collected for the determination of plasma concentrations of dronedarone and its metabolite N-desbutyl dronedarone. In each study period, samples are taken at pre-dose (0 h) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48, and 72 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects who voluntarily participate and provide written informed consent in accordance with Good Clinical Practice (GCP) guidelines.
2. Age ≥ 18 years.
3. Body weight ≥ 50.0 kg and body mass index (BMI) between 19.0 and 26.0 kg/m² (inclusive).
4. In good health as determined by comprehensive medical history, physical examination, and laboratory tests.
5. Able to comply with the study protocol and scheduled visits.

Exclusion Criteria:

1. Any clinically significant abnormalities in physical examination, vital signs, 12-lead ECG, cardiac ultrasound, or laboratory tests (including hematology, blood biochemistry, urinalysis, virology serology, and coagulation function).
2. History or presence of severe cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immune, dermatological, neurological, or psychiatric diseases. Specific exclusions include: renal insufficiency, heart failure, stroke, permanent atrial fibrillation, second- or third-degree atrioventricular block or sick sinus syndrome, bradycardia (heart rate < 50 bpm), prior amiodarone-associated hepatotoxicity or pulmonary toxicity, hypokalemia, hypomagnesemia, or family history of long QT syndrome.
3. History of specific allergies (e.g., asthma, urticaria, eczema), allergic constitution (allergy to two or more drugs or substances like milk/pollen), or known hypersensitivity to dronedarone, its components, or related compounds.
4. Major trauma or significant blood loss within 3 months prior to screening.
5. History of drug abuse within the past 5 years or positive urine drug screen.
6. Difficulty with blood sampling, needle phobia, or intolerance to venipuncture.
7. Positive alcohol breath test at screening.
8. Excessive alcohol consumption (>14 units per week; 1 unit = 285 mL beer, 25 mL spirits, or 100 mL wine) within 3 months prior to screening, or unwillingness to abstain from alcohol during the study.
9. Excessive consumption of tea, coffee, or caffeine-containing beverages (>8 cups per day; 1 cup = 250 mL) within 3 months prior to screening, or consumption of any alcohol, caffeine, or xanthine-rich products (e.g., coffee, strong tea, chocolate, cola, grapefruit) within 48 hours prior to dosing.
10. Inability to comply with a standardized diet, including food intolerance (e.g., to the standard meal), lactose intolerance, or dysphagia.
11. Smoking ≥5 cigarettes per day within 3 months prior to screening or unwillingness to refrain from smoking during the study.
12. Use of any medication (prescription, over-the-counter, herbal, or supplements) within 14 days prior to screening.
13. Use of any medication known to interact with dronedarone within 1 month prior to screening, including: QT-prolonging drugs, digoxin, calcium channel blockers, CYP2D6 substrates, potent CYP3A inhibitors, CYP3A inducers, statins, and narrow therapeutic index CYP3A substrates (e.g., dabigatran etexilate, warfarin).
14. Vaccination within 1 month prior to screening or planned vaccination during the study.
15. Participation in any other clinical trial within 3 months prior to screening.
16. Blood donation or significant blood loss (≥400 mL in total) within 3 months prior to screening.
17. Male subjects (or their partners) planning pregnancy from 2 weeks prior to screening until 3 months after study completion, or unwilling to use a medically acceptable non-pharmacological contraceptive method during the study.
18. Any other condition considered by the investigator as unsuitable for participation or voluntary withdrawal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours post-dose in each period
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 72 hours post-dose in each period
  plasma concentration-time curve from zero to the time of the last measurable time point t
Area under the plasma concentration versus time curve (AUC)0-∞ | 72 hours post-dose in each period
  area under the plasma concentration-time curve from zero to infinity

OTHER OUTCOMES:
maximum plasma concentration (tmax) | 72 hours post-dose in each period
  time to reach the maximum plasma concentration after drug administration (tmax)
Incidence of Treatment-Emergent Adverse Events | 24 days
  Collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital ＆ Institute (The Second Affiliated Hospital of Nanchang Medical College), Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No